CLINICAL TRIAL: NCT07220278
Title: Ongoing Dynamic Choice to Address HIV Treatment Interruption in Malawi (CHOICE)
Brief Title: Ongoing Dynamic Choice to Address HIV Treatment Interruption in Malawi
Acronym: CHOICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Partners in Hope, Inc. (Industry); Boston University (Other)
Responsible Party: Principal Investigator, Kathryn L. Dovel, PhD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH139452 (NIH); R01MH139452 (NIH)
Record Dates: First submitted 2025-10-15; First posted 2025-10-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: HIV
Keywords: client empowerment; HIV services; HIV treatment interruption; Malawi; eastern and southern Africa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHOICE (Experimental): The CHOICE intervention will provide long-term person-centered counseling + long-term, dynamic choice of DSD services to TI clients in Malawi over a 24-month period.
  Interventions: Behavioral: CHOICE
- Standard of Care (No Intervention): TI clients will be offered long-term person-centered counseling tailored to TI clients. The Malawi Ministry of Health adopted findings from previous trials and is incorporating short-term person-centered counseling into standard of care (SOC) for TI clients. This will be the SOC control condition.

INTERVENTIONS:
Behavioral: CHOICE — Routine HIV counselors will provide person-centered counseling and guide clients through a facilitated choice process to select DSDs and other support services routinely available to participating facilities. ART providers will review client preferences alongside client clinical assessments, resulting in a shared decision making of what DSD and support services is clinical safe and preferred for the client. Clients can change their preferred choice at any point throughout study enrollment. Ongoing, dynamic choice of available DSD models is a feasible and likely safe way to optimize the benefits of choice and provide responsive services for TI clients.
  Arms: CHOICE

SUMMARY:
Repeat and prolonged treatment interruption (TI) is common and the major threat to HIV epidemic control in eastern and southern Africa. The proposed project will test an innovative long-term dynamic choice intervention for ART clients experiencing TI in Malawi. Findings will provide essential information on how to improve sustained retention among TI client, a critical step to curbing the HIV epidemic. TI clients need long-term, responsive interventions. There are no one-size fits all intervention to support long-term care for TI clients because clients experience vastly different and changing barriers to care. While health facilities do have limited capacity for adding new services, existing services can be packaged differently to meet clients' needs.

Long-term, dynamic choice of services is one way to provide responsive services and promotes client ownership over care. The investigators propose to give TI clients long-term, dynamic choice of what services they receive and how they receive it (drawing from key building blocks of DSD). Long-term, dynamic choice puts clients in the driver's seat and may be the best practical strategy to provide long-term and responsive TI interventions that are tailored to clients' evolving life circumstances. Dynamic choice is frequently used for HIV prevention and family planning products, whereby clients select the type of health product that works best for them (i.e., condoms, injectables, etc.). Choice of these services is strongly associated with improved outcomes.

The goal of this clinical trial is to determine if CHOICE can improve outcomes in TI clients, compared to standard of care (SOC). Participants will be randomly assigned to either the CHOICE or SOC group, and follow them for 12 months. The primary outcome will be viral suppression at 12 months.

DETAILED DESCRIPTION:
Repeat and prolonged treatment interruption (TI) is common and the major threat to HIV epidemic control in eastern and southern Africa. The investigators define TI as >28 days late for last ART appointment. Each TI episode is associated with rapid viral load rebound and long-term decreases in CD4 count. Up to 46% of ART clients in the region experience TI in the first years after treatment initiation. 30-50% of clients returning from TI experience repeat TI <6 months after returning to care. TI and repeat TI account for the majority of HIV transmissions in Malawi. Strategies to provide ongoing support to TI clients are urgently needed.

Current TI services do not work in the long-term. The few evidence-based TI interventions that exist are extremely limited in duration (usually only ~1-3 intervention visits) and services offered (counseling alone or counseling + home-based initiation). Yet reasons for TI are different for each client and change over time. TI is rarely a one-time event. Short term interventions can improve return to care, but do not address repeat TI. The investigators' recent R01 (ENGAGE; R01MH122308-05, n=735) and BMGF (IDEAL; n=569) trials with men experiencing TI in Malawi show that short-term person-centered counseling + variations of short-term home-based ART dramatically improve return to care after TI (~96% re-initiated vs 67% in standard of care - SOC; p<0.001). But rates of continued ART engagement at 6-months after re-initiation (4-5 months after interventions completed) was unacceptably low (~64% were continuously in care without repeat TI vs 48% in SOC, p<0.001).

Recent trials found that clients with repeat TI had many unexpected and changing barriers that require long-term solutions. In-depth interviews with repeat TI clients in ENGAGE and IDEAL trials (n=67) showed that clients want long-term services responsive to their changing needs, and the ability to choose services.

TI clients need long-term, dynamic choice of differentiated service delivery (DSD) options. There are no one-size fits all interventions for TI clients because they experience vastly changing and different barriers to care, from distance to facility to lack of social support to limited HIV-related literacy. Ongoing person-centered counseling and choice of how services are delivered facilitates responsive services and promotes client ownership over care. Long-term and dynamic choice of DSD may be the best practical strategy to provide long-term, responsive TI interventions. There are no evidence-based dynamic choice interventions for TI clients.

The investigators piloted a novel intervention, called CHOICE, that provides person-centered counseling (building on the success of our prior trials) + ongoing, dynamic choice of DSD services to TI clients. The pilot (n=125) found that counseling + dynamic choice of DSD was feasible, acceptable, and showed signs of efficacy to reduce repeat TI (15% vs 50% at 3-months). A full trial is needed to test the impact on viral suppression long-term (at 12- and 24-months) and cost-effectiveness.

The investigators propose to evaluate CHOICE in a randomized control trial (RCT) with TI clients in Malawi. TI clients will receive person-centered counseling + ongoing, dynamic choice of how services are delivered (drawing on DSD models) over 24-months. Clients can combine multiple choices for service delivery at any given time to create personalized intervention packages. Choice of service delivery include: 1) ART dispensing intervals (1, 3, 6months), location of ART distribution (facility, home, or community), and peer mentorship (varying frequency and meeting location). Clients can adjust their choice at each ART visit or via hotline throughout study period. The investigators will compare CHOICE to SOC (1-3 counseling sessions + routine facility-based services - no choice available <6-months after TI. Specific aims are:

Aim 1. Test the effectiveness of CHOICE versus SOC on 12-month viral suppression among TI clients. The investigators will conduct an individually randomized trial at 12 health facilities (n=800 individuals). Primary outcome is viral suppression (<50copies/mL) at 12-months (study collected sample). Secondary outcomes are: presence of repeat TI, time to repeat TI, and ART coverage (days with ART in possession) across 24-months.

Aim 2: Systematically evaluate the implementation of CHOICE. The investigators will use mixed-methods to understand barriers, facilitators and needed improvements to HCW implementation of CHOICE, clients' ability to choose DSDs, and equity in intervention implementation and outcomes.

Aim 3. Estimate cost and cost-effectiveness of CHOICE. The investigators will use a micro-costing approach to estimate the distribution of care costs by study arm, differences between arms, and incremental cost effectiveness. The investigators will draw on patient-level resource use and unit costs developed from clinic and implementation financial data.

CHOICE will inform strategies for sustained retention among TI clients regionally and globally. The study is timely, of high-impact, and highly feasible within the Malawi health system and with our team. Malawi has a strong track record of implementing scientifically tested innovations into SOC that are high-impact and scalable, including several guidelines informed by our previous trials.

ELIGIBILITY:
Inclusion Criteria:

* 15 years of age or older
* living with HIV;
* initiated ART for the first time>3-months ago (i.e., not a new initiate);
* non-pregnant;
* experienced Treatment Interuptions during their most recent ARTappointment (>28 days late).

Exclusion Criteria:

* pregnant women because the ART/antenatal care (ANC) programs are integrated and require additional considerations and linkages with antenatal services.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of clients with viral suppression at 12-months (<1,000 copies/ML) | 12 months after enrollment
  Test the effectiveness of CHOICE versus SOC on 12-month viral suppression among TI clients. Primary outcome is viral suppression at 12-months (<1,000 copies/ML).

SECONDARY OUTCOMES:
Viral suppression at 24 months | 24 months after enrollment
  Number of participants with a viral load <1,000 copies/ML.
Advanced HIV at 12 and 24 months | at 12 and 24 months after enrollment
  Presence of HIV stage 3 or 4
ART re-initiation | 3 months after enrollment
  Percent of clients who re-initiate ART 3 months after enrollment
Repeat treatment interuption | 6, 12, and 24 months after enrollment.
  Proportion of clients who experience default (>28 days out of care) at any point in the first 6, 12, and 24 months after enrollment.
Adverse Events | Ongoing after enrollment to 24 months
  Presence of opportunistic infections or death after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L Dovel, PhD, Principal Investigator — University of California, Los Angeles; Augustine Choko, PhD, Principal Investigator — Partners in Hope, Inc.
Locations (1):
- Partners in Hope, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
An established repository will be used to ensure access that facilitates FAIRness (Findable, Accessible,Interoperable, and Re-usable) of the data. The metadata and other supporting documents will be submitted to the National Institute of Mental Health Data Archive (NDA) to facilitate scientific collaboration and data sharing.
  Per NDA guidelines, each participant will be assigned a global unique identifier (GUID) at trial enrollment, and informed consent will use appropriate language to convey data access and policies within NDA. All manuscripts and other dissemination materials will reference the Digital Object Identifier (DOI) associated with the appropriate data or document on NDA. Scientific data can also be found using standard indexing tools that optimize data locating via search engines. Keyword phrases for search engine optimization include: client empowerment for HIV services; HIV treatment interruption; Malawi; eastern and southern Africa.
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT07220278/Prot_SAP_000.pdf